CLINICAL TRIAL: NCT06856213
Title: TTCC-2022-02: A Phase II, Multicenter, Randomized Study of Cetuximab Plus/ Minus Weekly Paclitaxel After Progression To First-Line Pembrolizumab Plus Platinum-5FU in Subjects With Recurrent/Metastatic Squamous Cell Carcinoma of the Head and Neck (ERBIOTAX)
Brief Title: Study of Cetuximab Plus/Minus Weekly Paclitaxel After Progression To First-Line Pembrolizumab Plus Platinum-5FU in Subjects With Recurrent/Metastatic Squamous Cell Carcinoma of the Head and Neck.
Acronym: ERBIOTAX
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español de Tratamiento de Tumores de Cabeza y Cuello (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TTCC-2022-02; 2024-514953-31-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-06

CONDITIONS: Recurrent / Metastatic Head and Neck Squamous Cell Carcinoma
Keywords: Squamous Cell Carcinoma of the Head and Neck; SCCHN; Cetuximab; Paclitaxel
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab; Paclitaxel

STUDY DESIGN:
Intervention Model Description: Multi-center, open-label, randomized, non-comparative two-arm, phase 2 trial; Investigator Initiated Study (IIS).
  Patients will be randomized (2:1 ratio) to cetuximab + paclitaxel (ERBITAX) (Arm A) or to cetuximab monotherapy (Arm B).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARM A (Cetuximab+Paclitaxel) (Experimental): Cetuximab 400 mg/m2 initial dose followed by 250 mg/m2 + Paclitaxel 80mg/m2 (D1, D8 and D15 each 3-weeks cycle) for 4 cycles. Then, monotherapy maintenance with cetuximab at a dose of 500 mg/m2 will be administered biweekly (D1 and D15; Q4W) until disease progression or death, unacceptable toxicity or patient withdrawal of consent
  Interventions: Drug: Cetuximab; Drug: Paclitaxel
- ARM B (Cetuximab) (Experimental): Cetuximab 400 mg/m2 initial dose followed by 250 mg/m2 (D1, D8 and D15 each 3-weeks cycle) for 4 cycles. Then, maintenance with cetuximab at a dose of 500 mg/m2 will be administered biweekly (D1 and D15; Q4W) until disease progression or death, unacceptable toxicity or patient withdrawal of consent.
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Drug: Cetuximab — Cetuximab 250 mg/m2 will be administered as an intravenous infusion over 60 minutes. Cetuximab loading dose is 400 mg/m2 infusion and will be administered over 120 minutes. During maintenance, cetuximab at 500 mg/m2 will be administered as an intravenous infusion over 120 minutes.
Drug: Paclitaxel — Paclitaxel at a dose of 80 mg/m² will be administered after cetuximab as an intravenous infusion over 60 minutes weekly.
  Arms: ARM A (Cetuximab+Paclitaxel)

SUMMARY:
Squamous cell carcinoma of the head and neck (SCCHN) arises from epithelial cells and occurs in the oral cavity, pharynx and larynx. SCCHN is the seventh most common cancer worldwide with an annual incidence of approximately 90.000 cases per year in Europe.

Recurrent / metastatic SCCHN remains a grievous diagnosis and optimal treatment options after progression to first-line ICI treatment are not determined yet. Previous reports showed that cetuximab plus paclitaxel after progression to ICI therapy may have an enhanced activity as second line after ICI therapy ERBIOTAX is multi-center, open-label, randomized, non-comparative two-arm, phase 2 trial Investigator Initiated Study.

The primary study aims is to evaluate the efficacy of weekly cetuximab combined with paclitaxel (Arm A) or cetuximab monotherapy (Arm B) after progression to pembrolizumab plus platinum / 5-FU. The efficacy of treatment will be assessed through objective response rate (ORR).

Patients will be randomized in a 2:1 ratio to ERBITAX (cetuximab + paclitaxel) and cetuximab, respectively, assigning 2 patients to Arm A and 1 patient to Arm B out of 3 patients. No stratification for the randomization process is planned as this is a non-comparative study. A total of 65 evaluable patients will be included in the trial; 41 in Arm A and 24 in Arm B.

The main hypothesis is that treatment with the cetuximab +/- paclitaxel regimen maybe more effective after immune checkpoint inhibitors (ICI) failure in patients with recurrent/metastatic head and neck squamous cell carcinoma.

DETAILED DESCRIPTION:
1. Objectives

   Primary Objective

   -The study aims to evaluate the efficacy of weekly cetuximab combined with paclitaxel (Arm A) or cetuximab monotherapy (Arm B) after progression to pembrolizumab plus platinum / 5-FU. The efficacy of treatment will be assessed through objective response rate (ORR).

   Secondary Objectives
   * To evaluate clinical outcomes such as disease control rate (DCR), progression free survival (PFS), and overall survival (OS).
   * To evaluate the quality of life of patients with recurrent/metastatic head and neck squamous cell carcinoma treated with cetuximab and paclitaxel or cetuximab monotherapy.
   * To evaluate safety of the intended treatment regimen based on the frequency and severity of adverse events and Treatment-emergent adverse events (TEAEs) assessed by NCI CTCAE v5.0.

   Exploratory objectives
   * To evaluate the genomic/transcriptomic/proteomic alterations in baseline and on-treatment tumor samples.
   * To evaluate ctDNA dynamics between baseline and on-treatment plasma samples. Immunophenotyping of tumor samples.
2. Endpoints Primary Endpoint Confirmed objective response rate (ORR) according to RECIST V1.1 criteria Secondary Efficacy Endpoints

   * Disease Control Rate (DCR)

     . Median PFS
   * Median OS
   * Health-related quality of life (HRQoL), assessed through the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTC QLQ-C30) version 3, the head and neck specific module QLQ-H&N35 and EuroQol EQ-5D Secondary Safety Endpoints
   * Frequency and severity of adverse events and Treatment-related adverse events (TRAEs) assessed by NCI CTCAE v5.0
   * Rate of completion of C2D8, C4D8 and C6D8 of Cetuximab +/- Paclitaxel Exploratory endpoints
   * Presence of genomic/transcriptomic/proteomic alterations
   * ctDNA dynamics through study treatment
   * Immunophenotype of tumor and blood samples
3. Study Design The ERBIOTAX trial is a multicenter, open-label, randomized, non-comparative two-cohort, Phase II clinical trial of cetuximab either as monotherapy or in combination with paclitaxel in patients with SCCHN progressing on or after pembrolizumab plus platinum-based chemotherapy as first-line combination therapy. Additional details on the eligibility criteria of the study are found in protocol.

   The primary aim of the study is to evaluate the efficacy of weekly cetuximab combined with paclitaxel (Arm A) or cetuximab monotherapy (Arm B) after progression to pembrolizumab plus platinum / 5-FU. The efficacy of treatment will be assessed through ORR.

   The design includes a screening phase in which patient eligibility is addressed, a treatment phase with cetuximab, either as a single agent or combined with paclitaxel, and a follow-up phase.

   Signed informed consent form (ICF) will be obtained prior to the start of the specified screening window. Procedures conducted as part of the subject's routine clinical management (e.g., blood count determinations and imaging studies) prior to signing of ICF may be used for screening or for defining baseline data, provided these procedures are conducted as specified in the protocol.Patients will be randomized in a 2:1 ratio to ERBITAX and cetuximab, respectively.
4. Study population The trial will include 65 evaluable patients with recurrent/metastatic head and neck squamous cell carcinoma (41 in group A and 24 in group B).
5. Study Treatments

Patients will be randomized (2:1 ratio) to cetuximab + paclitaxel (ERBITAX) (Arm A) or to cetuximab monotherapy (Arm B). The complete schedule of treatment is detailed below:

ARM A: Cetuximab 400 mg/m2 initial dose followed by 250 mg/m2 + Paclitaxel 80mg/m2 (D1, D8 and D15 each 3-weeks cycle) for 4 cycles. Then, monotherapy maintenance with cetuximab at a dose of 500 mg/m2 will be administered biweekly (D1 and D15; Q4W) until disease progression or death, unacceptable toxicity or patient withdrawal of consent*.

ARM B: Cetuximab 400 mg/m2 initial dose followed by 250 mg/m2 (D1, D8 and D15 each 3-weeks cycle) for 4 cycles. Then, maintenance with cetuximab at a dose of 500 mg/m2 will be administered biweekly (D1 and D15; Q4W) until disease progression or death, unacceptable toxicity or patient withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

- Informed consent

1. Signed written and voluntary informed consent.
2. Patients must be willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.
3. Age > 18 years old. Disease characteristics
4. Have histologically confirmed diagnosis of head and neck squamous cell carcinoma.
5. The eligible primary tumor locations are oropharynx, oral cavity, hypopharynx, and larynx.
6. Known Human papillomavirus (HPV) status in oropharyngeal primaries and tested by p16 and/or HPV DNA testing by ISH or PCR. Local testing is acceptable.
7. Have confirmed disease progression per RECIST 1.1 on or after receiving platinum / 5-FU and pembrolizumab as first-line therapy for recurrent/metastatic disease. Patients must have measurable disease assessed by computed tomography (CT) scan or magnetic resonance imaging (MRI) based on RECIST 1.1 as assessed by the local site investigator/radiology. Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
8. All patients must provide a tumor biopsy obtained prior to the start of cetuximab +/- paclitaxel. A newly obtained biopsy -after progression to pembrolizumab + platinum-based chemotherapy - of a tumor lesion not previously irradiated for central biomarker analysis prior to start of study treatment is strongly preferred, but an archival sample may be acceptable upon discussion with the sponsor, if obtained in the prior 12 months.

   Note: Fine needle aspirate [FNA] is not adequate. Repeat samples may be required if adequate (quality and quantity) tissue is not provided. Formalin-fixed, paraffin embedded tissue blocks are preferred to slides

   Patient characteristics
9. Have a performance status of 0 or 1 on the ECOG Performance Scale
10. Patients must have adequate organ function as determined by the following. Screening labs should be performed within -7 days of treatment initiation:

    a. Hematology
    * Absolute neutrophils > 1.5 x 109/L
    * Platelets > 100 x 109/L
    * Hemoglobin > 90 g/L
    * Biochemistry
    * Bilirubin < 1.5 x upper limit of normal (ULN)
    * AST and ALT < 2.5 x ULN
    * Creatinine or measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤ 1.5xULN or ≥ 60 mL/min, respectively.

    Note: Hematology test should be obtained without transfusion or receipt of colony stimulating factors within 4 weeks prior to obtaining the sample.
11. Evidence of post-menopausal status, or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

    1. Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy).
    2. Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy).
12. Female subjects of childbearing potential should have a negative blood pregnancy test within 72 hours prior to receiving the first dose of study medication. A urine test can be considered if a blood test is not appropriate.
13. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile or abstain from heterosexual activity for the course of the study through 180 days after the last dose of study medication (6 months for paclitaxel). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for >1 year.

    Note: Abstinence is acceptable if this is the usual lifestyle and preferred method of contraception for the subject.
14. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 180 days after the last dose of study therapy (6 months for paclitaxel).

Note: Abstinence is acceptable if this is the usual lifestyle and preferred method of contraception for the subject.

Exclusion Criteria:

1. Patients with tumors of the head and neck region, arising from the nasopharynx, nasal cavity, paranasal sinuses, salivary glands, skin, unknown primary site.
2. Patients not treated or not progressing to pembrolizumab + platinum / 5-FU as the first line prior to their enrollment in the study. Progression to platinum / 5-FU plus pembrolizumab or other antiPD-(L)1 agents in combination with other immunotherapies including but not limited to other checkpoint regulatory monoclonal/bispecific antibodies such as anti CTLA-4, anti LAG-3 , anti TIGIT or anti TIM-3 may be allowed upon discussion with the sponsor.
3. Any previous treatment with paclitaxel and/or cetuximab in the recurrent or metastatic setting.
4. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.

   Note: Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging (using the identical imaging modality for each assessment, either MRI or CT scan) for at least 4 weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
5. Has a life expectancy of less than 3 months and/or has rapidly progressing disease (e.g. tumor bleeding, uncontrolled tumor pain) in the opinion of the treating investigator.
6. History of another primary malignancy, except for:

   1. Malignancy treated with curative intent and with no known active disease ≥3 years before the first dose of study drug and of low potential risk for recurrence,
   2. Adequately treated non-melanoma skin cancer without evidence of disease,
   3. Adequately treated carcinoma in situ without evidence of disease.
7. Any previous surgical treatment of the current cancer (except for a diagnostic biopsy) and no major surgery within 28 days prior to study treatment initiation. Performance of a tracheostomy or placement of a percutaneous gastrostomy tube within the 28 days prior to study treatment initiation will be allowed if the patient is clinically stable with no complications derived from those interventions.
8. Focal radiotherapy (RT) with palliative intent that is not completed 2 weeks prior to the first dose of Cetuximab +/- Paclitaxel.
9. History of allergic or hypersensitivity reactions to any study drugs or their excipients.
10. History of allogeneic organ transplant that requires therapeutic immunosuppression and the use of immunosuppressive agents within 28 days of study treatment initiation or a prior history of severe (grade 3 or 4) immune mediated toxicity from other immune therapy or grade ≥ 3 infusion reaction.
11. Any concurrent chemotherapy, biologic, immunologic or hormonal therapy for cancer treatment. Concurrent use of hormones for non-cancer-related conditions (eg, insulin for diabetes and hormone replacement therapy) is acceptable.
12. Current or prior use of immunosuppressive medication within 7 days prior to starting dosing. The following are exceptions to these criteria:

    1. Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra-articular injection).
    2. Adrenal replacement steroid > 10 mg daily prednisone equivalent are permitted in the absence of active autoimmune disease.
    3. Steroids as premedication for hypersensitivity reactions (eg, computed tomography scan premedication).
    4. < 10 mg prednisone or equivalent are permitted for the treatment of G1 IRAEs.
13. Any prior unresolved immune-related (ir) AE Grade > 2 not properly controlled as described in the exclusion criteria 14 and considered limiting according to physician criteria.
14. History of primary immune deficiency. History of organ transplant that requires use of immunosuppressive medications. Subjects who are human immunodeficiency (HIV) positive. Participants under definitive treatment for HIV (HAART) with undetectable viral load and >500 CD4+ T lymphocytes per μL at Screening Visit, are allowed.
15. History of stroke or transient ischemic attack within the previous 6 months.
16. Any of the following cardiac abnormalities:

    1. Unstable angina pectoris,
    2. Congestive heart failure ≥ NYHA Class 2,
    3. QTc (Fridericia formula) > 450 for males and > 470 ms for females,
    4. Known Left ventricular ejection fraction (LVEF) < 50,
    5. Unstable cardiac arrhythmia.
17. Pre-existing neuropathy ≥ Grade 2 per NCI CTCAE v5.0.
18. With history of interstitial lung disease, noninfectious pneumonitis, severe COPD, or uncontrolled lung diseases, including pulmonary fibrosis. However, specific cases may be allowed upon discussion with the sponsor.
19. Has a known history of or is positive for active hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (defined as HCV RNA [qualitative] is detected).

    Note: HBV DNA must be undetectable and HBsAg negative at Screening Visit. Active chronic hepatitis B on antiviral treatment with a negative viral load and preserved liver function is permitted upon consultation with the sponsor.

    Participants who have had definitive treatment for HCV are permitted if HCV RNA is undetectable at Screening Visit.
20. Female patients who are pregnant or breast-feeding.
21. Uncontrolled intercurrent illness including, but not limited to, ongoing or active clinically significant infection requiring parenteral antibiotics 2 weeks before treatment start,
22. Uncontrolled intercurrent psychiatric illness/social situations that would limit compliance with study requirements.
23. Any condition that, in the opinion of the Investigator, would interfere with evaluation of the study regimen or interpretation of patient safety or study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Confirmed objective response rate (ORR) according to RECIST V1.1 criteria | Throughout the study period, approximately 24 months
  Objective response rate (ORR) will be Assessed by the investigator through imaging follow-up (CT scan/MRI) using RECIST 1.1. This will be considered as the percentage/proportion of patients with confirmed complete response (CR) or partial response (PR) as their overall best response throughout the study period.
  Objective responses must be confirmed in a second CT scan performed 4 weeks later (+ 7 day window). Objective responses will be assessed locally by the investigator according to RECIST, version 1.1, and indicating the change in size of tumors as compared with baseline, at the first dose of study treatment.

SECONDARY OUTCOMES:
DCR (Disease Control Rate) | Throughout the study period, approximately in a time frame 6 months from the start of treatment
  Percentage/proportion of patients with complete response (CR) or partial response (PR), according to ORR definition for the trial, or maintained stable disease (SD) as their overall best response, assessed by imaging follow-up (CT scan/MRI) and RECIST 1.1 criteria. Stable disease should be maintained for at least 4 months to be considered as a DCR event.
Progression-free surviva (PFS) | Throughout the study period, at week 8 and every 12 weeks thereafter from start treatment for up to approximately 24 months
  Progression-free survival (PFS): Time from randomization to the date of confirmed PD according to RECIST 1.1. Patients alive and free of events at the date of the analysis will be censored at their last known tumor assessment. Patients who start a new treatment line without progression will be censored on the date of first dose of the subsequent anticancer treatment.
Overall survival (OS) | Throughout the study period, approximately 24 months from start treatment
  Overall survival (OS): defined as the time elapsed from randomization until death from any cause. We will assess the median OS, estimated by Kaplan-Meier. Patients alive and free of events at the date of the analysis will be censored at their last known contact. Survival will be assessed by recording patient status at each visit. Patients will be followed up for at least 2 years
Frequency and severity of adverse events and Treatment-related adverse events (TRAEs) | Throughout the study period, approximately a time frame of 2 years from start treatment
  Frequency and severity of adverse events and Treatment-related adverse events (TRAEs) assessed by NCI CTCAE v5.0 Adverse events (AE) assessment: type, frequency, outcome of adverse events and severe adverse events (SAEs). Actions taken regarding cetuximab and paclitaxel (i.e. treatment interruptions) will be recorded.
  Serious adverse events (SAEs) assessment: type, frequency, grade, outcome, relation with study treatment, all considering the total number and proportion based on the safety population.
  Treatment-related AEs: An event is assessed as related to study treatment when there is a reasonable possibility that study treatment caused the event. Reasonable possibility means there is evidence to suggest a causal relationship between study treatment and the event. This event is called a suspected adverse reaction. A suspected adverse reaction implies a lesser degree of certainty about causality than adverse reaction, which means any AE caused by a drug.
Health-related quality of life (HRQoL) | Throughout the study period, approximately a time frame of 2 years from start treatment
  Health-related quality of life (HRQoL), assessed through the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTC QLQ-C30) version 3, the head and neck specific module QLQ-H&N35 and EuroQol EQ-5D.
  These questionnaires ask questions in relation to physical, emotional, social aspects and in general the level of functionality of patients diagnosed with cancer in the last week after application.
  The scores range from 0 to 100. Higher scores indicate better functioning for the patients, except for symptoms scales, in which high scores indicate greaters symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Cabezas, M.D., Ph.D., Study Chair — Hospital San Carlos, Madrid; Marc Oliva, M.D., Ph.D., Study Chair — ICO-Hospitalet; Neus Basté, M.D, Study Chair — ICO-Badalona
Locations (11):
- Spain (11):
  - Instituto Catalán de Oncología - Hospital Duran i Reynals, Barcelona, Barcelona
  - Hospital Universitario Marqués de Valdecilla (Santander), Santander, Cantabria
  - Centro Oncológico de Galicia (La Coruña), A Coruña, La Coruña
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Universitario 12 de Octubre (Madrid), Madrid, Madrid
  - Hospital Infanta Leonor (Madrid), Vallecas, Madrid
  - Complejo Hospitalario de Navarra (Pamplona), Pamplona, Navarre
  - Complejo Hospitalario de Salamanca (Salamanca), Salamanca, Salamanca
  - Hospital Universitario de Canarias (La laguna), San Cristóbal de La Laguna, Santa Cruz de Tenerife
  - Hospital Universitario Virgen del Rocío (Sevilla), Seville, Sevilla
  - Hospital Universitario Virgen de Valme (Sevilla), Seville, Sevilla

IPD SHARING:
Plan to Share IPD: No